CLINICAL TRIAL: NCT07282405
Title: Validation of Alcohol Level Identification Using DRIVESC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-1470; Protocol Version 10/22/25 (Other: UW Madison); A561000 (Other: UW Madison)
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Driving Impaired
Keywords: drunk driving; alcohol
MeSH Terms: conditions — Driving Under the Influence | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Non-blinded three arm partial crossover
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alcohol Negative Day 1, Alcohol Negative Day 2 (Experimental): N = 6 participants, participants do not crossover
  Interventions: Diagnostic Test: DRIVESC
- Alcohol Negative Day 1, Alcohol Positive Day 2 (Experimental): N = 6-9 participants, prior to dosing day, participants must demonstrate 0.00 grams / 210 liter breath alcohol
  Interventions: Diagnostic Test: DRIVESC; Other: Alcohol
- Alcohol Positive Day 1, Alcohol Negative Day 2 (Experimental): N = 6-9 participants, prior to dosing day, participants must demonstrate 0.00 grams / 210 liter breath alcohol
  Interventions: Diagnostic Test: DRIVESC; Other: Alcohol

INTERVENTIONS:
Diagnostic Test: DRIVESC — Fitness to Drive Screening test battery and computer cognitive tests to assess divided attention, reaction time, and working memory
  Other Names: fitness to drive tests
Other: Alcohol — participants are dosed as part of the Wisconsin Basic Breath Examiner Specialist Training offered by the Chemical Testing Section (and not by the study team) over a one-hour period to a breath alcohol up to the legal limit of 0.08 percent grams/210 liter ethanol
  Other Names: ethanol
  Arms: Alcohol Negative Day 1, Alcohol Positive Day 2; Alcohol Positive Day 1, Alcohol Negative Day 2

SUMMARY:
This pilot study will evaluate the feasibility and acceptability of using a commercially available DRIVESC fitness-to-drive measurement tool to detect alcohol-induced impairment in healthy adult participants. The investigators hypothesize that DRIVESC can detect measurable changes in driving-related cognitive and motor performance across blood alcohol concentrations up to the U.S. per se legal limit of 0.08% g/210L ethanol. The study will enroll healthy adults aged 18-64 years (including both dosed and zero-alcohol arms) participating in the Wisconsin Breath Alcohol Examiner Specialist course, with each participant completing two study visits over two days.

DETAILED DESCRIPTION:
A total of 18-22 participants will be enrolled in this single-site partial crossover pilot study. Under the auspices of the Wisconsin Basic Breath Examiner Specialist training, participants will be dosed with alcohol on the first, second, or neither day of the three-day training.

This study design includes 6 double-alcohol-negative participants who will complete two days of alcohol-negative study tasks. The investigators will consider enrolling 12 alcohol-positive participants a success but are aiming to enroll 16 alcohol-positive participants. Alcohol-positive participants will complete two days of study tasks where one day is alcohol-negative and the other day is alcohol-positive. The order of positive-negative and negative-positive will be balanced. This range allows for flexibility in this feasibility study as study activities are scheduled in coordination with and around Chemical Testing Section training activities to minimize disruption to their educational tasks.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included in this study if they are trainees, observers, or instructors in the Wisconsin Basic Breath Examiner Specialist training program
* Meet the age requirements for their assigned study arm (18 years or older for non-drinking, 21 years or older for drinking), and
* Are able to provide informed consent.

Exclusion Criteria:

* Participants will be excluded from this study if they are unable to provide informed consent
* Do not meet the age requirements for their assigned study arm, or
* Are determined to be not suitable for participation due to other reasons at the discretion of the study team.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of Enrolled Participants who Complete all Scheduled Activities | through day 2
  Data will be recorded as completed vs not completed measurements or timepoints for each participant session.

SECONDARY OUTCOMES:
Within-Participant Change in DRIVESC Composite Score from Day 1 to Day 2: Non-Drinking Arm | through day 2
  The DRIVESC composite scoring is proprietary, but creates a single score representative of an individual's fitness to drive. It is calculated by combining the individual's performance on different cognitive and psychomotor assessments including measures of resilience, short-term memory recall, reaction ability, and completion of divided attention tasks. Scores range from 0-1 where 1 is the highest fitness to drive.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Barkholtz, PhD, Principal Investigator — UW School of Pharmacy
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No